CLINICAL TRIAL: NCT02972008
Title: Identification of Epigenetic Risk Factors for Ischemic Complication During the TAVR Procedure in the Elderly
Acronym: METHYSTROKE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_92; 2016-A01035-46 (Other: ID-RCB number); PHRCI_2015 (Other: PHRC number,DGOS)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Decline; Stroke
Keywords: Aortic stenosis; Transaortic valve replacement; stroke; Epigenetic
MeSH Terms: conditions — Cognitive Dysfunction; Stroke; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We compare the pre-operative leukocyte DNA methylation rate measured by the Luminometric Methylation Assay (LUMA) method in patients treated with TAVI and patients with constitutional von Willebrand factor (vWF) deficiency according to the presence or absence of at least one new cerebral ischemic lesion detected on postoperative cerebral MRI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cerebral Lesion: Patient over 70 years with severe aortic stenosis requiring percutaneous aortic valvular replacement (TAVI) having at least one new cerebral ischemic lesion on postoperative cerebral MRI
- No Cerebral Lesion: Patient over 70 years with severe aortic stenosis requiring percutaneous aortic valvular replacement (TAVI) with no cerebral ischemic lesion on postoperative cerebral MRI
- patients with constitutional von Willebrand factor (vWF) deficiency

SUMMARY:
Over the past ten years, the number of endovascular procedures has increased by 5% per year in Europe with the development of interventional cardiology, such as percutaneous coronary angioplasty, aortic valve replacements (TAVR), and vascular endoprosthesis.

The neurological lesions detected on cerebral MRI caused by these endovascular procedures are frequent with an incidence of about 30-70%. These events, although subclinical, have an impact on morbidity and mortality and especially on long-term cognitive decline.

TAVR is the reference treatment for symptomatic elderly patients with stenosis of the aortic valve, considered by a multidisciplinary "Heart Team" as at high surgical risk due to comorbidities, age and high perioperative risk scores ( Euroscore 2 and STS scores). Despite the net clinical benefit, an increase of silent neurological events was detected on post-procedural cerebral MRI with an incidence of approximately 70%.

The epigenetic involvement in the occurrence of ischemic cerebral lesions is still largely unknown. Epigenetic mechanisms, such as DNA methylation, can be associated with aging processes and modulate the risk of developing cerebrovascular pathologies. They are likely to provide new biomarkers that predict the risk of brain damage.

Hypomethylation of leukocyte DNA is directly related to atherosclerosis in humans. This hypomethylation of DNA would represent an easily measurable marker reflecting the presence and progression of atherosclerosis. Because atherosclerotic lesions often precede the clinical manifestation of ischemic cardiovascular disease, such as ischemic heart disease and stroke, DNA hypomethylation could be used to identify individuals at risk for cerebrovascular events.

The investigator hypothesize that hypomethylation of leukocyte DNA can predict the risk of developing new ischemic brain lesions especially after a TAVI procedure.

DETAILED DESCRIPTION:
This is a french multicenter prospective cohort study. Patients with severe symptomatic aortic stenosis referred for a TAVI procedure to the cardiology departments of the university hospitals of Lille, Caen, Amiens and the Pitié-Salpêtrière hospital (APHP) are analyzed for inclusion in this prospective study. The cases are selected after a discussion between the members of the local TAVI "Heart Team" (cardiologists, cardiac surgeons, anesthetists), as recommended by the guidelines of the European Society of Cardiology. Written consent is obtained in accordance with international recommendations for clinical research (Helsinki Declaration). Participation in the study is proposed to patients during preoperative consultation.

The collection of clinical data, including postoperative cerebral MRI, is collected prospectively during hospitalization and during the clinical visit to each institution at one year. An evaluation of cognitive function is performed by a mini-mental state (MMS) the day before the TAVI intervention and then at 1 year. The study ends after the last evaluation. A cerebral MRI is performed within 1-3 days after the TAVI procedure to detect new cerebral ischemic lesions (emboli).

Blood samples will be taken during the patient's stay: the day before TAVI, during the procedure and after the TAVI procedure at day 1 and day 4.

The follow-up visit to 1 year will be conducted by cardiologists or cardiac surgeons with an evaluation of the cognitive function by the mini-mental state (MMS).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 70 years with severe aortic stenosis requiring percutaneous aortic valve replacement (TAVI)

Exclusion Criteria:

* Patient contraindicated for the TAVI procedure
* Patient with a pace-maker
* Patient with contra-indication for cerebral MRI
* Ongoing cancer
* Patient already involved in therapeutic research
* Major persons under protection of justice.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 70 years with severe aortic stenosis requiring percutaneous aortic valve replacement (TAVI)
Sampling Method: Probability Sample
Enrollment: 542 (Estimated)
Dates: Start 2017-03-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pre-operative leukocyte DNA methylation rate | Within one week after the procedure
  This rate will be measured by the LUMA method in patients treated with TAVI according to the presence of at least one new cerebral ischemic lesion and/or microbleeds cerebral lesion appearing on post-procedural MRI

SECONDARY OUTCOMES:
Variation of the leukocyte DNA methylation rate during the TAVI procedure | At time between the pre (day-1) and postprocedural (day 1) samples
  This rate will be measured by the LINE-1 method in all patients
Pre-operative leukocyte DNA methylation rate (stroke/TIA) | One day before the procedure and within one week after the procedure
  This rate will be measured by the LUMA method in patients treated with TAVI according to the presence of a neurological deficit (stroke, transient ischemic attack)
Mortality | At 1 year after procedure
  The mortality in patients treated with TAVI according to the presence of at least one new micro-ischemic cerebral lesion and/or one new microbleeds cerebral lesion detected on postoperative cerebral MRI and / or postprocedural ischemic stroke / TIA
MMSE score variation | At day-1 before TAVI procedure, at 6 months and at 1 year after procedure
  The MMSE score variation is compared according to the presence or not of at least one new micro-ischemic cerebral lesion and/or one new microbleeds cerebral lesion
Change of EQ-5D questionnaire | At day-1 before TAVI procedure, at 6 months and at 1 year after procedure
  The evolution of quality of life is compared to the occurrence of new cerebral events one new micro-ischemic cerebral lesion and/or one new microbleeds cerebral lesion
Change of modified Rankin Scale (mRS) | At day-1 before TAVI procedure, at 6 months and at 1 year after procedure
  The MRS (measure degree of disability- troke) is compared to the occurrence of new cerebral events one new micro-ischemic cerebral lesion and/or one new microbleeds cerebral lesion
Change of National Institutes of Health Stroke Scale (NIHSS) | At day-1 before TAVI procedure, at 6 months and at 1 year after procedure
  TheNIHSS (quantify the impairment caused by a stroke) is compared to the occurrence of new cerebral events one new micro-ischemic cerebral lesion and/or one new microbleeds cerebral lesion
Clinical and Biological predictors of new cerebral events | At day-1 before TAVI procedure, at 6 months and at 1 year after procedure
  The clinical (measured before the procedure) and biological characteristics of the patients (measured before the procedure and after the procedure) and of the peri-procedural parameters associated with the occurrence of new events detected on post-procedural MRI (new ischemic and/or new microbleeds cerebral lesion appearing on post-procedural MRI)
Hemostasis predictors of new cerebral events | At day-1 before TAVI procedure, at 6 months and at 1 year after procedure
  Hemostasis parameters (measured before the procedure and after the procedure) including Willebrand factor parameters associated with the occurrence of new events detected on postoperative MRI (new ischemic and/or new microbleeds cerebral lesion)
Number of complications in peri-procedural according to VARC-2 criteria | Within one week after the procedure
  Evaluation of multi criteria according to the Valve academic Research Consortium (VARC-2)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Debry, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital cardiologie, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghanem A, Kocurek J, Sinning JM, Wagner M, Becker BV, Vogel M, Schroder T, Wolfsgruber S, Vasa-Nicotera M, Hammerstingl C, Schwab JO, Thomas D, Werner N, Grube E, Nickenig G, Muller A. Cognitive trajectory after transcatheter aortic valve implantation. Circ Cardiovasc Interv. 2013 Dec;6(6):615-24. doi: 10.1161/CIRCINTERVENTIONS.112.000429. Epub 2013 Oct 15. PMID 24129642
- [Background] Kahlert P, Knipp SC, Schlamann M, Thielmann M, Al-Rashid F, Weber M, Johansson U, Wendt D, Jakob HG, Forsting M, Sack S, Erbel R, Eggebrecht H. Silent and apparent cerebral ischemia after percutaneous transfemoral aortic valve implantation: a diffusion-weighted magnetic resonance imaging study. Circulation. 2010 Feb 23;121(7):870-8. doi: 10.1161/CIRCULATIONAHA.109.855866. PMID 20177005
- [Background] Bjornsson HT, Sigurdsson MI, Fallin MD, Irizarry RA, Aspelund T, Cui H, Yu W, Rongione MA, Ekstrom TJ, Harris TB, Launer LJ, Eiriksdottir G, Leppert MF, Sapienza C, Gudnason V, Feinberg AP. Intra-individual change over time in DNA methylation with familial clustering. JAMA. 2008 Jun 25;299(24):2877-83. doi: 10.1001/jama.299.24.2877. PMID 18577732
- [Background] Baccarelli A, Wright R, Bollati V, Litonjua A, Zanobetti A, Tarantini L, Sparrow D, Vokonas P, Schwartz J. Ischemic heart disease and stroke in relation to blood DNA methylation. Epidemiology. 2010 Nov;21(6):819-28. doi: 10.1097/EDE.0b013e3181f20457. PMID 20805753
- [Background] Van Belle E, Juthier F, Susen S, Vincentelli A, Iung B, Dallongeville J, Eltchaninoff H, Laskar M, Leprince P, Lievre M, Banfi C, Auffray JL, Delhaye C, Donzeau-Gouge P, Chevreul K, Fajadet J, Leguerrier A, Prat A, Gilard M, Teiger E; FRANCE 2 Investigators. Postprocedural aortic regurgitation in balloon-expandable and self-expandable transcatheter aortic valve replacement procedures: analysis of predictors and impact on long-term mortality: insights from the FRANCE2 Registry. Circulation. 2014 Apr 1;129(13):1415-27. doi: 10.1161/CIRCULATIONAHA.113.002677. Epub 2014 Feb 24. PMID 24566199
- [Background] Gilard M, Eltchaninoff H, Iung B, Donzeau-Gouge P, Chevreul K, Fajadet J, Leprince P, Leguerrier A, Lievre M, Prat A, Teiger E, Lefevre T, Himbert D, Tchetche D, Carrie D, Albat B, Cribier A, Rioufol G, Sudre A, Blanchard D, Collet F, Dos Santos P, Meneveau N, Tirouvanziam A, Caussin C, Guyon P, Boschat J, Le Breton H, Collart F, Houel R, Delpine S, Souteyrand G, Favereau X, Ohlmann P, Doisy V, Grollier G, Gommeaux A, Claudel JP, Bourlon F, Bertrand B, Van Belle E, Laskar M; FRANCE 2 Investigators. Registry of transcatheter aortic-valve implantation in high-risk patients. N Engl J Med. 2012 May 3;366(18):1705-15. doi: 10.1056/NEJMoa1114705. PMID 22551129
- [Result] Van Belle E, Debry N, Vincent F, Kuchcinski G, Cordonnier C, Rauch A, Robin E, Lassalle F, Pontana F, Delhaye C, Schurtz G, JeanPierre E, Rousse N, Casari C, Spillemaeker H, Porouchani S, Pamart T, Denimal T, Neiger X, Verdier B, Puy L, Cosenza A, Juthier F, Richardson M, Bretzner M, Dallongeville J, Labreuche J, Mazighi M, Dupont-Prado A, Staels B, Lenting PJ, Susen S. Cerebral Microbleeds During Transcatheter Aortic Valve Replacement: A Prospective Magnetic Resonance Imaging Cohort. Circulation. 2022 Aug 2;146(5):383-397. doi: 10.1161/CIRCULATIONAHA.121.057145. Epub 2022 Jun 20. PMID 35722876